CLINICAL TRIAL: NCT06940869
Title: Network to Understand Reproductive Rheumatology Registry
Acronym: NURTURE
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00117179
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Rheumatic Diseases; Pregnancy Related; Pregnancy Interest; Reproductive Health; Autoimmune Diseases
MeSH Terms: conditions — Rheumatic Diseases; Autoimmune Diseases | interventions — Family Planning Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NURTURE Registry — To improve pregnancy and birth outcomes for women with rheumatic diseases and to understand risk factors associated with poor pregnancy outcomes.
  Other Names: Women with rheumatic/autoimmune diseases who are pregnant or planning pregnancy

SUMMARY:
The purpose of the NURTURE Registry is to enroll those who are pregnant and/or potentially capable of pregnancy. Participants will complete patient-reported surveys at enrollment and periodically prior to conception, during pregnancy, and following the completion of the study pregnancy. The study rheumatologist will provide the patient's diagnosis and record rheumatic disease activity at each clinic visit. Medication use, vital signs, and routine laboratory assessments will be collected throughout this period. Pregnancy, maternal, and infant outcomes will be obtained through the electronic medical record and from patient-reported surveys. This Registry will provide a rich data repository for research to improve pregnancy and birth outcomes for women with rheumatic diseases and will be used in on-going and future research to better understand the risk factors that are associated with poor pregnancy outcomes, including preterm birth, intrauterine growth restriction, and preeclampsia, as well as the effects of medication on disease management in pregnancy. Infant outcomes, medications, provider care, pregnancy planning, and social determinants of health on pregnancy and pregnancy outcomes will also be collected.

The majority of the information collected in NURTURE, such as labs, disease activity, and medications, PRO's will originate from the EHR. Upon consent, participants will complete an enrollment survey that will include relevant patient reported measures. No study visits outside of routine care will occur. Participants may also complete a yearly survey about their reproductive health journey.

The registry will be ongoing and will include periodic analysis of clinical data within this protocol. Additional analysis will be covered under seperate IRB approved protocols. Enrollment in the registry does not significantly increase the risk for a patient.

DETAILED DESCRIPTION:
The purpose of the NURTURE Registry is to obtain information on those who are pregnant and/or potentially capable of pregnancy. This Registry will provide a rich data repository for research to improve pregnancy and birth outcomes for women with rheumatic diseases and will be used in on-going and future research to better understand the risk factors that are associated with poor pregnancy outcomes, including preterm birth, intrauterine growth restriction, and preeclampsia, as well as the effects of medication on disease management in pregnancy. Infant outcomes, medications, provider care, pregnancy planning, and social determinants of health on pregnancy and pregnancy outcomes will also be collected.

Participation in NURTURE will be seamless with routine patient care. Any patient with a rheumatic disease seen by a participating site study provider as part routine care, and who could potentially become pregnant (females between the ages of 12 and 55), or who is currently pregnant, will be invited to participate in NURTURE. Participants will complete patient-reported surveys at enrollment and periodically prior to conception, during pregnancy, and following the completion of the study pregnancy. The study rheumatologist will provide the patient's diagnosis and record rheumatic disease activity at each clinic visit. Medication use, vital signs, and laboratory assessments will be collected as part of standard clinical care vistis and used in this registry. Pregnancy, maternal, and infant outcomes will be obtained through the electronic medical record and from patient-reported surveys.

Prior to or at each standard of care (non-study, routine) visit, the patient will complete routine clinical questionnaires.

This is a natural-history study and will not include medications, laboratory testing, or procedures outside of the standard of care. Management of the rheumatologic disease will be directed based on patient needs by the local rheumatologist and obstetrician.

Enrollment in the registry will not dictate specific therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of an automimmune or rheumatic condition determined by health care provider.
2. Age 12-55 who are capable of pregnancy (currently pregnant or planning a pregnancy).
3. A patient who receives their care in the Duke Health System.
4. Capable of providing informed consent.

Exclusion Criteria:

1. Unable to provide informed consent.

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Capable of pregnancy
Study Population: Currently pregnant or desire to become pregnant and have an autoimmune or rheumatic condition.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Edinburgh post-partum depression scale | up to 20 years
  Depression at entry in NURTURE defined by the Edinburgh Postnatal Depression Scale (EPDS) score ≥10 indicating minor depression.

SECONDARY OUTCOMES:
Readiness for Pregnancy | up to 20 years
  We will explore the effect size of the HOP-STEP Intervention on 'personally-ready and 'medically-ready' pregnancies by comparing women who did and did not receive the HOP-STEP Intervention.
  "Medically ready" will be defined as <1g of proteinuria, no rheumatic teratogens at conception, and continuing pregnancy compatible SLE medications after conception.
  "Personally ready" will be defined as a planned pregnancy based on a London Measure of Unplanned Pregnancy (LMUP) score ≥10.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Clowse, Principal Investigator — Professor of Medicine, Duke University Health System
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No